CLINICAL TRIAL: NCT02386449
Title: A Randomized, Controlled, Parallel Group, Assessor-Blinded Study To Compare The Efficacy, Tolerability, And Safety Of Oral Sodium Picosulfate (PicoPrep®) Versus Oral Mannitol and Bisacodyl, For Colon Cleansing In Colonoscopy Preparation Of Adult Outpatients
Brief Title: A Study Comparing Picoprep With Mannitol and Bisacodyl for Colon Cleansing in Preparation for Colonoscopy
Acronym: CLEAR PREP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 000180
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — picosulfate sodium; Magnesium Oxide; Citric Acid; Mannitol; Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Picoprep (Experimental): sodium picosulfate, magnesium oxide and citric acid
  Interventions: Drug: sodium picosulfate, magnesium oxide and citric acid (Picoprep®)
- Mannitol and Bisacodyl (Active Comparator)
  Interventions: Drug: mannitol; Drug: Bisacodyl

INTERVENTIONS:
Drug: sodium picosulfate, magnesium oxide and citric acid (Picoprep®)
  Arms: Picoprep
Drug: mannitol
  Arms: Mannitol and Bisacodyl
Drug: Bisacodyl
  Arms: Mannitol and Bisacodyl

SUMMARY:
This is a randomized, controlled, parallel group, assessor-blinded study to compare two colon cleansing preparations for colonoscopy. Subjects meeting all inclusion and exclusion criteria will be randomized and assigned to one of two study groups: Group I (PicoPrep) or Group II (Mannitol). In Group I, subjects will take one sachet of PicoPrep on the day before colonoscopy, and another sachet on the day of colonoscopy. In Group II, subjects will take Bisacodyl on the day before colonoscopy, and Mannitol on the day of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 60 years
* Subjects scheduled for an elective colonoscopy
* Women of child-bearing potential using at least one highly effective contraceptive method
* Subjects able to understand all instructions
* Informed consent signed

Exclusion Criteria:

* Hypersensitivity to active ingredients
* Female participants pregnant or with a positive blood pregnancy test
* Acute surgical abdomen
* Previous colorectal surgery
* Gastrointestinal (GI) surgery
* GI diseases, active inflammatory bowel disease, colon disease
* Ascites/hepatic cirrhosis, cardiac disease, advanced pulmonary or renal disease
* Use of laxatives or antidiarrheal agents 72 hours prior to screening
* Significant alterations in laboratory values or other diseases that could interfere with the results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects classified as success (Aronchick scale) | At visit 2 (day 1 of colonoscopy)
  Defined as excellent or good according to the Aronchick scale

SECONDARY OUTCOMES:
Percentage of subjects classified as success (Ottawa scale) | At visit 2 (day 1 of colonoscopy)
  Defined as excellent, good or fair according to the Ottawa scale
Aggregate Tolerability Score (Colonoscopy Preparation Subject Tolerability Questionnaire) | At visit 2 (day 1 of colonoscopy)
  As assessed by a Colonoscopy Preparation Subject Tolerability Questionnaire
Subject satisfaction (Likert scale) | At visit 2 (day 1 of colonoscopy)
  As assessed by a subject survey using a 3 point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (there may be other sites in this country), São Paulo, Brazil